CLINICAL TRIAL: NCT00490841
Title: A Clinical Trial to Assess the Safety and Efficacy of the RX Herculink(R) Elite(TM) Renal Stent System for the Treatment of Suboptimal Post-procedural Percutaneous Transluminal Angioplasty (PTA) in de Novo or Restenotic Renal Artery Stenoses in Patients With Uncontrolled Hypertension.
Brief Title: The HERCULES Trial - A Safety and Effectiveness Study of the Herculink Elite Renal Stent to Treat Renal Artery Stenosis
Acronym: HERCULES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-102
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Renal Artery Obstruction; Hypertension, Renal
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RX Herculink Elite (Experimental): To evaluate the safety and effectiveness of the RX Herculink Elite Renal Stent System in the treatment of suboptimal post-procedural percutaneous transluminal angioplasty (PTA) of atherosclerotic de novo or restenotic renal artery stenosis in patients with uncontrolled hypertension.
  Interventions: Device: Herculink Elite Renal Stent System

INTERVENTIONS:
Device: Herculink Elite Renal Stent System — This is a prospective, non-randomized, single arm, multi-center study to evaluate the safety and effectiveness of the RX Herculink Elite Renal Stent System in patients with sub-optimal renal PTA results in de novo or restenotic renal artery lesions. Patients who satisfy the inclusion/exclusion criteria will be enrolled at sites in the United States. Patients will have follow up visits for evaluation.

SUMMARY:
The purpose of this study is to determine whether the Herculink Elite Renal Stent System is safe and effective in the treatment of renal artery stenosis in patients with less than optimal angioplasty results and uncontrolled hypertension.

CAUTION: The Herculink Elite Renal Stent System Is An Investigational Device. Limited by Federal (U.S.) Law to Investigational Use Only.

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of the RX Herculink Elite Renal Stent System in the treatment of suboptimal post-procedural percutaneous transluminal angioplasty (PTA) of atherosclerotic de novo or restenotic renal artery stenosis in patients with uncontrolled hypertension.

CAUTION: The Herculink Elite Renal Stent System Is An Investigational Device. Limited by Federal (U.S.) Law to Investigational Use Only.

ELIGIBILITY:
General Clinical Inclusion Criteria:

* Subject is ≥18 years of age.
* Subject and subject's physician agree to have the subject return for all required contact following study enrollment.
* Subject has been informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site.
* Subject is a candidate for renal artery stenting.
* Subject has uncontrolled systolic hypertension (systolic Blood Pressure[SBP] ≥140 mmHg), or uncontrolled diastolic hypertension (diastolic BP [DBP] ≥90 mmHg), or a combination of both in the presence of at least two (2) or more antihypertensive medications.
* Subject has a baseline serum Creatinine of <2.5mg/dl

Angiographic Inclusion Criteria

* Subject has either unilateral or bilateral de novo or restenotic after Percutaneous Transluminal Angioplasty (PTA) (in-stent restenosis excluded) atherosclerotic lesion(s). If bilateral lesions are to be treated, the most severe lesion must be successfully treated without complications before progressing to treat the second lesion. Treatment of bilateral lesions is to occur in the same procedural event.
* Renal stenosis must be visually estimated to be ≥60% by angiography.
* Subject has a suboptimal PTA result, defined as one of the following:

  * ≥50% residual stenosis
  * 10 mm Hg mean gradient or 20 mm Hg peak systolic gradient across the target lesion
  * A flow-limiting dissection (NHLBI grade D) or TIMI flow <3
* Renal stenosis must be visually estimated to be within 10 mm of the aortic renal border by angiography.
* Target vessel reference diameter must be visually estimated to be ≥4mm and ≤7mm by angiography
* Target lesion length must be visually estimated to be ≤15mm (including dissection) by angiography.
* Expected ability to deliver the stent to the lesion (absence of excessive tortuosity or calcification).
* Expected ability to fully expand the stent.

Clinical Exclusion Criteria

* Subject has known hypersensitivity or contraindication to cobalt chromium or standard intraprocedure anticoagulant(s); subject has sensitivity to contrast which cannot be adequately pre-treated with medication.
* Subject has known allergy or contraindication to clopidogrel (Plavix) or aspirin.
* Subject has known bleeding disorder or hypercoagulable disorder, or will refuse blood transfusions.
* Subject has suffered a gastrointestinal (GI) bleed within 30 days before the index procedure that would interfere with antiplatelet therapy.
* Subject has renal insufficiency defined as serum Creatinine >2.5 mg/dl.
* Subject has any immunosuppressive disorder, access site infection, or acute systemic infection due to any cause.
* Subject has other medical illnesses (e.g., cancer, end-stage congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation, or is associated with a life expectancy of less than three years.
* Subject has any medical illnesses that would make them unlikely to respond to treatment (e.g., sickle cell nephropathy/sickle cell disease, scleroderma, arteriolar nephrosclerosis, hemolytic-uremic syndrome and vasculitis).
* Subject has had a Q-wave MI within 30 days before index procedure.
* Subject has had a stroke or TIA within 30 days before index procedure.
* Subject has a history of congestive heart failure and has a previously documented LVEF ≤25%.
* Subject is normotensive or has adequate control of hypertension (SBP <140 mmHg and DBP <90 mm Hg) utilizing diet control and/or medication regimen involving only one antihypertensive medication.
* Subject has acute thrombophlebitis or deep vein thrombosis.
* Subject is actively participating in another drug or device trial and has not completed the required protocol follow-up period. Subject may be enrolled only once in this study (Protocol # 05-102) and may not participate in any other clinical trial during the follow-up period.
* Subject is unable to understand and cooperate with study procedures or provide informed consent.
* Subject is unable to return for follow-up visits (distance, etc).
* Subject is pregnant.
* Subject has undergone vascular surgery (CABG, AAA repair, AF bypass) and has not fully recovered from the effects of surgery (<3 months).
* Subject has planned staged treatment of bilateral renal artery stenosis.
* Subject has had prior surgical intervention to the target artery, or has undergone previous stent placement in the target lesion.
* Target lesion is located in a transplanted kidney.
* Kidney to be treated is <8 cm as determined by duplex ultrasound report, CTA report, or MRA report within 180 days before procedure. If kidney size is documented by more than one method, e.g. CTA and ultrasound, and one of the methods is duplex ultrasound, the kidney size as documented by duplex ultrasound shall be used to determine study eligibility.
* Subject has planned additional ancillary procedure(s) during renal stenting procedure.

Angiographic Exclusion Criteria

* Subject has a lesion segment, including dissection, >15 mm in length.
* Requirement for >1 stent to treat full length of lesion and dissection.
* Target lesion has a total (100%) occlusion.
* Evidence of thrombus or mobile filling defect in the target lesion or vessel.
* Subject has co-existing aneurysmal or occlusive disease of the abdominal aorta requiring surgical reconstruction during the follow-up period.
* Target lesion is non-atherosclerotic (fibromuscular dysplasia).
* Subject artery has patent bifurcation within 10 mm of ostium that might be covered by placement of a stent.
* The target lesion is within the artery of a solitary functioning kidney or, the subject has a contralateral totally occluded renal artery.
* For planned treatment of bilateral lesions: the more critical lesion, i.e. lesion with the greater stenosis (which should be treated first), is either treated unsuccessfully or requires a bailout procedure. (NOTE: Less critical lesion is excluded at this point.)
* Subject has any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe.
* The target lesion is densely calcified and will not yield during balloon dilation.
* Subject has had recent change in renal function after unrelated catheter or surgical procedure with the clinical stigmata of atheroemboli syndrome (i.e., livedo reticularis: non-occlusive mesenteric ischemia; digital gangrene; progressive renal insufficiency without other identifiable etiology).
* Subject has an accessory renal artery that has >50% stenosis. Accessory renal arteries may not be stented as part of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bates, MD, Study Director — CAMC Health System; Stephen Textor, MD, Study Director — Mayo Clinic; Michael Jaff, DO, Study Director — Vascular Diagnostic Laboratory; Timothy Sullivan, MD, Study Director — Heart Hospital of SD; Andrew Blum, MD, Study Director — Midwest Heart Foundation
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Jaff MR, Bates M, Sullivan T, Popma J, Gao X, Zaugg M, Verta P; HERCULES Investigators. Significant reduction in systolic blood pressure following renal artery stenting in patients with uncontrolled hypertension: results from the HERCULES trial. Catheter Cardiovasc Interv. 2012 Sep 1;80(3):343-50. doi: 10.1002/ccd.24449. Epub 2012 Jun 27. PMID 22511402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects admitted for percutaneous renal artery revascularization were considered for enrollment at sites throughout the USA. Dates of enrollment: August 31, 2007 through October 02, 2009.
Pre-assignment Details: Subjects required to have documented uncontrolled hypertension (SBP at least 140 mmHg or DBP at least 90 mmHg, or both) in the presence of at least two (2) or more antihypertensive medications, all clinical eligibility criteria had to have been met and sujects had to sign the informed consent form. Intent to treat (ITT) population.
Period: Overall Study
Arm/Group | RX Herculink Elite
Started | 202
Completed | 189
Not Completed | 13
Not completed — Death | 5
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — 30 day f/u, only non-study stent used | 3

BASELINE CHARACTERISTICS:
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 163
Age Continuous [Mean (Standard Deviation); unit: years] | 72.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 202

OUTCOME MEASURES:

1. Primary Outcome: Binary Restenosis Rate
Description: Determined by duplex ultrasound or angiogram. Reported as the percentage of participants with occurance of binary restenosis.
Time Frame: 9 months
Population: Subject total reflects those who were evaluable at the time of analysis. The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician. Only a certain number of patients were required to have angiographic follow-up to provide this endpoint information.
Measure: Number (95% Confidence Interval); unit: Percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 178
Number analyzed (Lesions) | 209
Percentage of lesions | 10.5 [NA to 14.7] — One-sided confidence interval was computed for this endpoint, lower bound is not provided.
Statistical Analysis 1: Comparison: RX Herculink Elite; objective is to demonstrate the binary restenosis rate at 9 months is < 28.6% OPC. Assumptions for the primary endpoint analysis: * H0: Restenosis Rate ≥ 28.6% * HA: Restenosis Rate < 28.6% * Assumed binary restenosis rate = 20% * Power = 80% * One-sided type I error = 5% With the above assumptions, 161 samples would be required. To account for approximately 20% lost to follow-up rate, 202 subjects will be enrolled in the study. The sample size calculation was performed using PASS 2005; Test type: Superiority or Other; p < 0.0001, 1-sided exact binomial test

2. Secondary Outcome: Death for Any Reason
Time Frame: 30 days
Population: Non-Hierarchical Subject Counts, Per Subject Analysis (Intent-to-Treat Population). The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 201
percentage of participants | 0.5 [0.0 to 2.7]

3. Secondary Outcome: Ipsilateral Nephrectomy
Description: Ipsilateral: Situated on or affecting the same side as treated. Nephrectomy: Removal of the affected kidney
Time Frame: 30 days
Population: intention to treat (ITT). The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RX Herculink Elite: Subjects recieving the RX Herculink Elite
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 201
percentage of participants | 0 [0.0 to 1.8]

4. Secondary Outcome: Embolic Events Resulting in Kidney Damage
Description: Percentage of participants with an embolic event resulting in kidney damage.
Time Frame: 30 days
Population: The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 201
Percentage of participants | 1.0 [0.1 to 3.5]

5. Secondary Outcome: Event Free Rate of Clinically Indicated Target Lesion Revascularization (TLR)
Description: Event Free percentage: Defined as percentage of participants free from this event.
Time Frame: 9 months
Population: as for outcome 4
Measure: Number; unit: Event Free Percentage
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 201
Event Free Percentage | 96.9

6. Secondary Outcome: 9 Month Blood Pressure (Systolic)
Description: As compared to baseline (pre-procedure). Blood pressure measurements at 9 months.
Time Frame: Baseline (Pre-Procedure) and 9 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 173
mmHg
  9 month Systolic Blood Pressure | 145.3 [142.1 to 148.5]
  Baseline (Pre-Procedure) Systolic Blood Pressure | 162.3 [159.8 to 164.9]

7. Secondary Outcome: 9 Month Blood Pressure (Diastolic)
Description: As compared to baseline. See Population description.
Time Frame: 9 months and baseline
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 173
mmHg
  9 month Diastolic Blood Pressure | 75.4 [73.6 to 77.1]
  Baseline Diastolic Blood Pressure | 77.7 [76.1 to 79.3]

8. Secondary Outcome: Acute Device Success
Description: Acute device success is defined as, on a per device basis, the achievement of successful delivery of the assigned device(s)as intended to the designated location.
Time Frame: From beginning of index procedure to end of index proceedure.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: Devices
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 202
Number analyzed (Devices) | 247
percentage of devices | 96.0 [92.7 to 98.0]

9. Secondary Outcome: Acute Procedure Success
Description: Attainment of a final result of < 30% residual stenosis, as determined by the Angiographic Core Lab.
Time Frame: From beginning of index proceedure to end of index proceedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 202
Number analyzed (Lesions) | 240
percentage of participants | 99.2 [97.0 to 99.9]

10. Secondary Outcome: Acute Clinical Success
Description: Procedure success without Major Adverse Events (MAE)or access site event requiring surgical or percutaneous intervention prior to hospital discharge.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: From beginning of index proceedure to end of index proceedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 201
percentage of participants | 98 [95 to 99.5]

11. Secondary Outcome: Primary Patency
Description: Defined as <60% stenosis without prior re-intervention, as determined by duplex ultrasound or angiogram.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Subject total reflects those who were evaluable at the time of analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 178
Number analyzed (Lesions) | 209
percentage of participants | 88 [82.9 to 92.1]

12. Secondary Outcome: Secondary Patency Rate of <60% Stenosis of the Target Lesion
Description: As determined by duplex ultrasound or angiography regardless of PTA, stenting, or bypass since index procedure. Rate reported as a percentage of participants with this condition.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Subject total reflects those who were evaluable at the time of analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 177
Number analyzed (Lesions) | 208
percentage of participants | 95.2 [91.3 to 97.7]

13. Secondary Outcome: 9 Month Anti-hypertensive Medication In-take, 1 Medication
Description: Number of Anti-Hypertensive Medications taken-baseline compared to follow up, Per Subject Analysis (Intent-to-Treat Population), reported as the percentage of participants using the number of medications indicated.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Patients with baseline Anti-Hypertensive medication intake equal to 1 medication: 0.5%
Measure: Number; unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 174
percentage of participants | 4.6

14. Secondary Outcome: 9 Month Anti-hypertensive Medication In-take, 2 Medications
Description: Number of Anti-Hypertensive Medications taken-baseline compared to follow up, Per Subject Analysis (Intent-to-Treat Population)), reported as the percentage of participants using the number of medications indicated.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Patients with baseline Anti-Hypertensive medication intake equal to 2 medications: 29.2%
Measure: Number; unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 174
percentage of participants | 29.3

15. Secondary Outcome: 9 Month Anti-hypertensive Medication In-take, 3 Medications
Description: as for outcome 14
Time Frame: 9 months
Population: Patients with baseline Anti-Hypertensive medication intake equal to 3 Medications: 30.7%
Measure: Number; unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 174
percentage of participants | 28.2

16. Secondary Outcome: 9 mo in Anti-hypertensive Medication In-take, ≥ 4 Medications
Description: Number of Anti-Hypertensive Medications taken at follow up compared to baseline, Per Subject Analysis (Intent-to-Treat Population)), reported as the percentage of participants using the number of medications indicated.
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Patients with baseline Anti-Hypertensive medication intake equal to or greater than 4 Medications: 39.6%
Measure: Number; unit: percentage of participants
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 174
percentage of participants | 37.4

17. Secondary Outcome: Renal Function (Measured by sCr)
Description: sCR= Serum Creatinine, per subject analysis. ITT. Renal function (measured by sCr) @ baseline: 1.2mg/dL (1.2, 1.3).
  The analysis population at clinical follow-up visits may have changed due to early termination from the study by the patient or physician.
Time Frame: 9 months
Population: Subject total reflects those who were evaluable at the time of analysis.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | RX Herculink Elite
Number analyzed (Participants) | 167
mg/dL | 1.3 (0.6) [1.2 to 1.4]

ADVERSE EVENTS:
Time Frame: Post-procedure through 312 days
Description: Organ systems designations were chosen to match Abbott Categories coding as closely as possible and may differ from other coding systems.
Arm/Group | RX Herculink Elite
Serious Adverse Events (participants affected / at risk) | 83/199
Other Adverse Events (participants affected / at risk) | 145/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RX Herculink Elite (N=199)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) — Access site complication
Pseudoaneurysm (Surgical and medical procedures) | 1 (1) — Access Site Complication
Blood Dyscrasia (Blood and lymphatic system disorders) | 6 (6) — Anemia
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Acute Myocardial Infarction (Cardiac disorders) | 5 (6)
Angina (Cardiac disorders) | 5 (5) — Cardiac/Hemodynamic
Arrhythmias (Bradycardia & Tachycardia) (Cardiac disorders) | 9 (11) — Cardiac/Hemodynamic
Cardiac Arrest (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Cardiomyopathy (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Chest Pain (Cardiac disorders) | 2 (2) — Cardiac/Hemodynamic
Congestive Heart Failure (Cardiac disorders) | 7 (7) — Cardiac/Hemodynamic
Hypertension Exacerbation (Cardiac disorders) | 7 (8) — Cardiac/Hemodynamic
Hypotension (Cardiac disorders) | 2 (2) — Cardiac/Hemodynamic
Pacemaker Issue (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Unstable Angina (Cardiac disorders) | 6 (7) — Cardiac/Hemodynamic
Appendicitis (Gastrointestinal disorders) | 1 (1) — Gastrointestinal
Diarrhea (Gastrointestinal disorders) | 2 (2) — Gastrointestinal
Digestive Disorder (Gastrointestinal disorders) | 4 (4) — Gastrointestinal
Diverticulitis (Gastrointestinal disorders) | 1 (1) — Gastrointestinal
Nausea (Gastrointestinal disorders) | 2 (2) — Gastrointestinal
Pyloric Channel Ulcer (Gastrointestinal disorders) | 2 (2) — Gastrointestinal
Vomiting (Gastrointestinal disorders) | 2 (2) — Gastrointestinal
Joint/Bone (Infections and infestations) | 2 (3) — Infection
Urinary Tract Infection (Infections and infestations) | 1 (1) — Infection
Viral, Bacterial and Fungal Infections (Infections and infestations) | 4 (4) — Infection
Electrolyte Imbalance (Metabolism and nutrition disorders) | 6 (6) — Metabolic
Back Pain (General disorders) | 2 (2) — Miscellaneous
Edema (Non Pulmonary) (General disorders) | 1 (1) — Miscellaneous
Joint Pain (General disorders) | 3 (3) — Miscellaneous
Joint/Bone (General disorders) | 1 (1) — Miscellaneous
Lightheadedness/Dizziness (General disorders) | 2 (2) — Miscellaneous
Medication Side Effect (General disorders) | 1 (1) — Miscellaneous
Myalgia (General disorders) | 1 (1) — Miscellaneous
Pain (General disorders) | 1 (1) — Miscellaneous
Syncope (General disorders) | 4 (4) — Miscellaneous
Trauma (General disorders) | 3 (3) — Miscellaneous
Vision Disturbance (General disorders) | 1 (1) — Miscellaneous
Weight Gain/Loss (General disorders) | 1 (1) — Miscellaneous
Neuropathy (Nervous system disorders) | 1 (1) — Neurological
Stroke/Cerebral Vascular Accident (Nervous system disorders) | 4 (4) — Neurological
Transient Ischemic Attack (Nervous system disorders) | 1 (1) — Neurological
GI Bleed (Blood and lymphatic system disorders) | 5 (5) — Non-Access Site Bleeding
Retroperitoneal Bleed (Blood and lymphatic system disorders) | 2 (2) — Non-Access Site Bleeding
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary/Respiratory
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Pulmonary/Respiratory
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Pulmonary/Respiratory
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary/Respiratory
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Pulmonary/Respiratory
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary/Respiratory
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Pulmonary/Respiratory
Creatinine Increase (Renal and urinary disorders) | 2 (2) — Renal
Cysts/Stones (Renal and urinary disorders) | 1 (1) — Renal
Insufficiency (Renal and urinary disorders) | 4 (4) — Renal
Renal Failure (Renal and urinary disorders) | 2 (3) — Renal
Claudication (Vascular disorders) | 2 (2) — Vascular
Ischemia (Vascular disorders) | 1 (1) — Vascular
Restenosis (Vascular disorders) | 15 (16) — Vascular
Stenosis (Vascular disorders) | 16 (21) — Vascular
Thrombosis (Vascular disorders) | 2 (2) — Vascular
Total Occlusion (Vascular disorders) | 2 (2) — Vascular
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RX Herculink Elite (N=199)
Bleeding (Surgical and medical procedures) | 12 (12) — Access Site Complication
Hematoma (Surgical and medical procedures) | 19 (20) — Access Site Complication
Hypertention Exacerbation (Cardiac disorders) | 27 (28) — Cardiac/Hemodynamic
Digestive Disorder (Gastrointestinal disorders) | 12 (12) — Gastrointestinal
Nausea (Gastrointestinal disorders) | 14 (15) — Gastrointestinal
Urinary Tract Infection (Infections and infestations) | 12 (13) — Infection
Back Pain (General disorders) | 22 (24) — Miscellaneous
Fatigue/Weakness (General disorders) | 11 (12) — Miscellaneous
Joint Pain (General disorders) | 11 (11) — Miscellaneous
Lightheadedness/Dizziness (General disorders) | 15 (16) — Miscellaneous
Myalgia (General disorders) | 11 (14) — Miscellaneous
Pain (General disorders) | 13 (14) — Miscellaneous

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days